CLINICAL TRIAL: NCT03347643
Title: Randomized Double-blind Clinical Trial to Evaluate the Effectiveness of Transcranial Direct Current Stimulation (tDCS) on Internet Game Addiction
Brief Title: The Effectiveness of tDCS on Internet Game Addiction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Seok Choi, Clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30-2017-10
Record Dates: First submitted 2017-11-13; First posted 2017-11-20 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Addiction; Internet Gaming Disorder
Keywords: Internet game addiction; Internet gaming disorder; transcranial direct current stimulation; response inhibition; craving; cue reactivity
MeSH Terms: conditions — Behavior, Addictive; Internet Addiction Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Patients with internet gaming disorder will be randomly allocated into 1) actual real stimulation with tDCS group, and 2) sham stimulation with tDCS group.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS with real stimulation (Active Comparator): A total of 25 patients will be allocated into active comparator with real stimulation with tDCS.
  Interventions: Device: tDCS with real stimulation
- tDCS with sham stimulation (Sham Comparator): A total of 25 patients will be allocated into sham comparator with sham stimulation with tDCS.
  Interventions: Device: tDCS with sham stimulation

INTERVENTIONS:
Device: tDCS with real stimulation — tDCS is a non-invasive brain stimulation. Real stimulation includes 2mA current for 20 minutes per session. Two sessions a day for 5 consecutive days (Total: 10 sessions) will be applied.
  Arms: tDCS with real stimulation
Device: tDCS with sham stimulation — Sham stimulation includes 0mA current for 20 minutes per session. Two sessions a day for 5 consecutive days (Total: 10 sessions) will be applied.
  Arms: tDCS with sham stimulation

SUMMARY:
In this study, the investigators aimed to investigate the effect of transcranial direct current stimulation (tDCS) on clinical status of Internet game addiction. The clinical status of Internet game addiction includes severity of addiction symptom, subjective craving for gaming, response inhibition and cue reactivity. The investigators hypothesized that real stimulation with tDCS on the dorsolateral prefrontal cortex will have higher effectiveness on severity of addiction symptom, subjective craving for gaming, response inhibition and cue reactivity rather than sham stimulation with tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Internet gaming disorder based on diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders (DSM)-5.

Exclusion Criteria:

* History of seizure
* History of significant head injury
* Mental retardation
* Schizophrenia
* History of stroke

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Young Internet Addiction Test (Y-IAT) | baseline
  The Y-IAT is rated on a five-point scale. Total scores for all 20 items range from 20 to 100.
Young Internet Addiction Test (Y-IAT) | 1 week
  The Y-IAT is rated on a five-point scale. Total scores for all 20 items range from 20 to 100.
Young Internet Addiction Test (Y-IAT) | 5 week
  The Y-IAT is rated on a five-point scale. Total scores for all 20 items range from 20 to 100.
Young Internet Addiction Test (Y-IAT) | 25 week
  The Y-IAT is rated on a five-point scale. Total scores for all 20 items range from 20 to 100.

SECONDARY OUTCOMES:
Direction error and successful stop ratio in the Stop signal task | baseline, 5 weeks, 25 weeks
  The stop signal task is a neurocognitive task for assessing response inhibition.
Barratt impulsiveness scale-11 | baseline, 5 weeks, 25 weeks
  Barratt impulsiveness scale-11 is a self-report questionnaire consisting of 30 items. Each question has a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/always). This scale scores three subscales: attentional impulsiveness, motor impulsiveness, and nonplanning impulsiveness. The total score ranges from 30 to 120 and higher scores indicate greater impulsivity.
Anti-saccade error rate in the attentional bias task | baseline, 5 weeks, 25 weeks
  The attentional bias task is measured by anti-saccade task using eye-tracking analysis for assessing attentional bias on Internet gaming stimuli.
Late positive potential in the cue reactivity event-related potential | baseline, 5 weeks, 25 weeks
  Event-related potential measures with cue reactivity task
Visual analogue scale | baseline, 1 week, 5 weeks, 25 weeks
  Subjective craving for Internet gaming ranging from 0 to 10. Higher score represents higher craving for gaming.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Seok Choi, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JY, Jang JH, Choi AR, Chung SJ, Kim B, Park M, Oh S, Jung MH, Choi JS. Neuromodulatory Effect of Transcranial Direct Current Stimulation on Resting-State EEG Activity in Internet Gaming Disorder: A Randomized, Double-Blind, Sham-Controlled Parallel Group Trial. Cereb Cortex Commun. 2021 Jan 4;2(1):tgaa095. doi: 10.1093/texcom/tgaa095. eCollection 2021. PMID 34296150